CLINICAL TRIAL: NCT03867357
Title: Intramuscular Mechanisms of Androgen Deprivation-related Sarcopenia
Status: Completed | Type: Observational
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: 1653
Record Dates: First submitted 2019-02-26; First posted 2019-03-08 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Prostate Cancer; Androgen Deprivation Therapy
Keywords: Androgen deprivation therapy; Prostate cancer; Sarcopenia
MeSH Terms: conditions — Prostatic Neoplasms; Sarcopenia | interventions — Gonadotropin-Releasing Hormone; Goserelin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, muscle samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: GnRH agonist — Zoladex is a gonadotropin-releasing hormone agonist, or GnRH-A. It is an implant that is injected under the skin (subcutaneously). The implant gradually dissolves and releases the drug over the time between injections. There are two dosages of Zoladex: Zoladex 10.8 mg, which is injected once every 3 months, and Zoladex 3.6 mg, which is injected once a month.
  Other Names: Zoladex, Goserelin

SUMMARY:
Prostate cancer (PCa) is the most common cancer among men and is even more common in the military and veteran population. For patients with advanced prostate cancer, the most common treatment includes lowering the levels of the hormone testosterone as much as possible. This is called "androgen deprivation therapy" or "ADT". Unfortunately, ADT also causes patients to be fatigued, weak and to loose muscle. This is often referred to as "sarcopenia" and it leads to falls, poor quality of life and higher risk of death. Currently, there is no treatment for sarcopenia because the investigators do not understand the mechanisms that cause it. The mitochondria is the part of the cells responsible for providing energy to muscles but to this date the investigators do not know if it is affected in prostate cancer patients with sarcopenia due to ADT.

The overall goal of this proposal is to establish if the mitochondria is responsible for sarcopenia in patients with prostate cancer receiving ADT. The investigators will measure mitochondrial function, muscle mass and strength, and feelings of fatigue and quality of life in patients with prostate cancer before starting and after 6 months of ADT.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most common cancer among men. Androgen deprivation therapy (ADT) is the standard treatment for advanced and metastatic PCa and nearly 400,000 men remain on androgen deprivation therapy (ADT) for advanced PCa in the U.S. Unfortunately, ADT also induces a decrease in muscle mass and function, known as sarcopenia, a condition that leads to decreased endurance, increased fatigue, falls, poor health-related quality of life (HR-QOL) and increased mortality. The mechanisms underlying the development of ADT-induced sarcopenia are incompletely understood and remain a significant barrier to the development of therapies for this condition. Mitochondria play an essential role in generating the adenosine triphosphate (ATP) needed for muscle contraction and abnormalities in mitochondria function have been reported in animal models of sarcopenia. The extent to which mitochondrial dysfunction mediates ADT-induced sarcopenia and muscle dysfunction is not known.

The overall goal of this proposal is to establish the role of mitochondrial dysfunction on ADT-induced sarcopenia in patients with PCa. The investigators hypothesize that ADT in men with PCa will induce mitochondrial dysfunction leading to sarcopenia.

Improving scientific understanding of the mechanisms underlying sarcopenia following ADT will enable investigators to develop new treatments and novel biomarkers for this disease. Given that there are no available therapies for sarcopenia, this is clinically very relevant. The near-term impact of this proposal will be to elucidate the extent to which mitochondrial dysfunction mediates the development of sarcopenia in veterans and non-veterans with prostate cancer undergoing ADT, and to evaluate the potential for these measurements at baseline to serve as early predictors of disease. The outcomes that will be directly attributed to the results of the proposed research include baseline and changes in muscle mass and performance, in-vivo and ex-vivo mitochondrial function, and patient reported outcomes (PROs) including fatigue and HR-QOL. The investigators expect that these efforts will have a major impact on the goal of reducing morbidity associated with prostate cancer, and improving HR-QOL by filling the gap in the knowledge of the mechanisms causing ADT-induced sarcopenia in PCa. The mechanisms identified in this grant will be the target of future interventional clinical trials.

The proposed project will address one of the PCRP overarching challenges and focus areas: "Survivorship including psychosocial impact on the patient". If the investigators prove the hypothesis that mitochondrial dysfunction plays a significant role in the development of sarcopenia, fatigue and poor HR-QOL in veterans and non-veterans with prostate cancer, the multidisciplinary team that has been assembled will build on these findings and test interventions currently undergoing clinical development to target mitochondria dysfunction in this population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically, cytologically, or image based documented advanced or metastatic PCa initiating ADT with expected continuous treatment for a minimum of 6 months and willing/able to provide informed consent.
* Willing and able to provide written informed consent prior to screening.

Exclusion Criteria:

* Liver disease (AST or ALT equal or more than 3x normal levels);
* Renal failure (creatinine equal or more than 2.5 mg/dL);
* Untreated thyroid disease, class III-IV CHF, AIDS;
* Other cancer diagnosed within the past five years other than non-melanoma skin cancer;
* Severe COPD requiring use of home O2;
* Chronic, uncontrolled hypertension as judged by the Investigator (i.e., Baseline SBP >150 mm Hg, DBP >90 mm Hg) or a SBP > 150 mm Hg or DBP > 95 mm Hg at the time of screening or baseline;
* An active, uncontrolled infection or cardiovascular disease including a recent myocardial infarction (MI), cerebrovascular accident (CVA), arrhythmias or unstable angina (< 6 months);
* Uncontrolled diabetes mellitus (as defined by a HbA1c equal or more than 9%);
* Underlying muscular or neuromuscular disorder or neurologic deficit contributing to sarcopenia;
* Enrolled in a clinical trial involving an investigational product or non-approved use of a drug/device or concurrently enrolled in medical research not scientifically or medically compatible with this study;
* Current use (within one month) of testosterone, high dose steroids (20mg of prednisone/day for more than 1 month), or megestrol treatment for cancer within the previous 3 months;
* Previous treatment with ADT other than oral anti-androgen at initiation of ADT;
* Metal implants in the right limbs (non-MRI compatible metal stents, titanium pins/markers, etc.) or implanted cardiac pacemaker or other implanted non-MRI compatible cardiac device (e.g., stent);
* A history of vascular problems (DVT, etc.)

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male Veteran patients presenting with advanced or metastatic PCa eligible for ADT in the Urology clinic at the Veterans Affairs Puget Sound Health Care System.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Lean body mass (LBM) change | Baseline to 3 months
  Changes in LBM (kg) measured by X-ray densitometry (DEXA).
Lean body mass (LBM) change | Baseline to 6 months
  Changes in LBM (kg) measured by X-ray densitometry (DEXA).

SECONDARY OUTCOMES:
Body composition change | Baseline to 6 months
  Lean body mass and fat mass (kg) measured by dual energy x-ray absorptiometry (DEXA)
Muscle strength change | Baseline to 6 months
  Hand grip strength (kg)
Muscle strength change | Baseline to 6 months
  Stair climb power (seconds)
Muscle thickness change | Baseline to 6 months
  Changes in muscle thickness by Ultrasound
Aerobic capacity change | Baseline to 6 months
  VO2 max
Daily physical activity change | Baseline to 6 months
  Actigraphy
Skeletal muscle mitochondrial function (in vivo) | Baseline to 6 months
  Magnetic resonance spectroscopy (MRS)
Skeletal muscle mitochondrial function (ex vivo) | Baseline to 6 months
  Oxygen consumption rate (OCR)
Quality-of-life change | Baseline to 6 months
  EORTC Quality of Life Questionnaire (EORTC QLQ-C30)
Quality-of-life change | Baseline to 6 months
  Expanded Prostate Cancer Index Composite (EPIC) questionnaire
Quality-of-life change | Baseline to 6 months
  Functional Assessment of Cancer Therapy-Prostate questionnaire

OTHER OUTCOMES:
Degree of androgen deprivation | Baseline to 6 months
  Total and free testosterone levels in blood draw samples

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Garcia, MD, PhD, Principal Investigator — Veterans Affairs Puget Sound Health Care System, University of Washington
Locations (1):
- Veterans Affairs Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shanely RA, Zwetsloot KA, Triplett NT, Meaney MP, Farris GE, Nieman DC. Human skeletal muscle biopsy procedures using the modified Bergstrom technique. J Vis Exp. 2014 Sep 10;(91):51812. doi: 10.3791/51812. PMID 25285722

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT03867357/Prot_SAP_000.pdf